CLINICAL TRIAL: NCT06267742
Title: Clinical Trial to Evaluate Early Sepsis Indicator Monocyte Distribution Width (MDW) for Early Detection of Sepsis or Developing Sepsis
Brief Title: Clinical Trial to Evaluate MDW for Early Detection of Sepsis
Status: Active, not recruiting | Type: Observational
Sponsor: Beckman Coulter, Inc. (Industry)
Collaborators: Peking Union Medical College Hospital (Other); West China Hospital (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: CHN097
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Blood Cell Count

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Diagnostic Test: Complete Blood Count (CBC) with Differential — CBC with Differential including Monocyte Distribution Width (MDW)

SUMMARY:
This study is intended to clinically verify Monocyte Distribution Width (MDW) parameter of DxH 900 Hematology Analyzer for use in early detection and risk assessment of sepsis, severe sepsis, and septic shock in critically ill patients in Emergency Department (ED). This study is also aimed to provide study supporting data for the product to be marketed in China.

DETAILED DESCRIPTION:
To verify the clinical performance of MDW parameter in detection of sepsis through a multicenter, prospective study of adults undergoing complete blood count with differential ("CBC with differential") in the ED.

To clarify the cutoff 20.0 established in the pivotal trial. The cutoff was established for the objective of achieving the highest sensitivity at the optimal specificity level. Patients whose MDW value is higher than the cutoff will be identified as sepsis patients and those whose MDW value is equal to or lower than the cutoff are non-sepsis patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (18-89 years) presenting to ED.
* CBC with Differential performed upon presentation as part of standard of care.
* Subject scheduled for at least 12 hours follow-up during ED (or inpatient, if admitted to the hospital) visit
* Signed the informed consent form

Exclusion Criteria:

* Subjects previously enrolled in this study (i.e., re-enrollment to this study is not allowed).
* The subject is discharged from the hospital within 12 hours after ED visit

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of any race and ethnicity can be enrolled to this study. Patients with a prior chronic immunosuppressive disease and subjects with hematological malignancy can also be enrolled. This study requires at least 250 sepsis subjects and 1,100 non-sepsis subjects.
Sampling Method: Non-Probability Sample
Enrollment: 2200 (Estimated)
Dates: Start 2022-06-23 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
sensitivity, specificity | 2022.3-2024.3
  sensitivity (percentage of patients with sepsis correctly identified), specificity (percentage of non-sepsis patients correctly identified) according to Sepsis-2

CONTACTS AND LOCATIONS:
Overall Officials: DONG LI, MS, Study Director — BECKMAN COULTER
Locations (3):
- China (3):
  - Peking Union Medical College Hospital, Beijing
  - West China Hospital, Sichuan University, Chengdu
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou

IPD SHARING:
Plan to Share IPD: No